CLINICAL TRIAL: NCT05447715
Title: Fruquintinib Sequential BEV+FOLFIRI vs. BEV+FOLFIRI Sequential Fruquintinib in the Treatment of Metastatic Colorectal Cancer That Has Failed Previous Fluorouracil/Oxaliplatin Therapy
Brief Title: Fruquintinib Sequential BEV+FOLFIRI vs. BEV+FOLFIRI Sequential Fruquintinib in Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Weijian Guo (Other)
Responsible Party: Sponsor-Investigator, Weijian Guo, Chief physician, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FBIRI
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; Fruquintinib; bevacizumab (BEV); FOLFIRI; second-line treatment; third-line treatment
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fruquintinib sequential BEV+FOLFIRI (Other)
  Interventions: Drug: Fruquintinib
- BEV+FOLFIRI sequential fruquintinib (Other)
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib sequential BEV+FOLFIRI vs. BEV+FOLFIRI sequential fruquintinib in the treatment of metastatic colorectal cancer that has failed previous fluorouracil/oxaliplatin therapy

SUMMARY:
This is a prospective, open, multicenter, randomized controlled phase II study designed to observe the difference of efficacy, adverse events and quality of life between second-line and third-line application of Fruquintinib in patients with metastatic colorectal cancer. The study will evaluate PFS, ORR, OS and safety.

DETAILED DESCRIPTION:
A maximum of 134 patients with metastatic colorectal cancer who had previously failed to receive fluorouracil/oxaliplatin were included in the study. The patients were randomly divided into two groups according to the ratio of 1:1 and given different medication regiments. Stratified factors included left and right colorectal cancer, tumor RAS gene status, and first-line use of bevacizumab. Specific grouping and medication regimen are as follows:

Second-line treatment group (F-C group) : After enrollment, patients were given Fruquintinib 5 mg/d orally for 21 consecutive days with 7 days of rest, with a cycle of 28 days. Use drugs until the disease progresses or toxicity is intolerable, and then carry out third-line treatment. BEV+FOLFIRI was administered in the third line. Third-line medication until disease progression or toxicity becomes intolerable.

Third-line application group (C-F group) : After enrollment, patients were treated with BEV+FOLFIRI until disease progression or toxicity intolerance, and third-line treatment was carried out after progression. Fruquintinib was given in the third line of treatment, specifically: Fruquintinib 5 mg/d orally for 21 consecutive days, followed by 7 days of rest, with a cycle of 28 days. Third-line medication until disease progression or toxicity becomes intolerable.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent;
2. Be 18 or older;
3. patients with metastatic colorectal adenocarcinoma confirmed by histopathology or cytopathology;
4. Failure of first-line oxaliplatin combined with fluorouracil (combined with or without targeted therapy);
5. With one or more measurable lesions, the longest diameter determined by spiral CT scan should be at least 10 mm, and the longest diameter determined by conventional CT scan should be at least 20 mm (efficacy evaluation criteria for solid tumors, namely RECIST criteria, version 1.1);
6. Eastern Oncology Collaboration group (ECOG) General status score 0 or 1;
7. The expected survival time is more than 3 months;
8. Hematopoietic function, liver and kidney function should meet the following criteria within 7 days before screening:

   Absolute neutrophil count ≥ 1.5x109 /L; Hemoglobin ≥ 9.0g/dL; Platelet count ≥ 80 x109 /L; Total bilirubin ≤1.5 times normal upper limit (ULN); Alanine aminotransferase and aspartate aminotransferase ≤ 2.5 x ULN; Alkaline phosphatase ≤ 3 x ULN; Serum creatinine ≤1.5 x ULN;
9. Men, women of reproductive age (postmenopausal women must have been in menopause for at least 12 months to be considered infertile), and their partners voluntarily used contraceptive methods that the investigator considered effective during treatment and for at least six months after the last study drug was taken.

Exclusion Criteria:

Subjects who meet any of the following criteria will not be enrolled:

1. BRAF V600E mutation confirmed by histological or blood ctDNA gene test;
2. Heavy tumor load (such as liver tumor accounting for more than 50% of the liver volume, or a single tumor lesion with a diameter of more than 5 cm, or chest tightness, shortness of breath and other symptoms, lung metastasis that has affected respiratory function);
3. First-line treatment with irinotecan;
4. The patient has ascites or peritoneal metastasis;
5. Uncontrolled pleural effusion;
6. There is a risk of bleeding, such as a large surgical operation within one month or a small needle biopsy within two weeks; There was active gastrointestinal bleeding. Severe unhealed wounds; Hereditary bleeding tendency or coagulopathy.
7. History of gastrointestinal perforation or abdominal abscess within 6 months prior to enrollment.
8. Uncontrolled hypertension (systolic blood pressure & GT; 150mmHg and/or diastolic pressure > 100mmHg), clinically significant cardiovascular disease, such as symptomatic coronary artery disease or myocardial ischemia (myocardial infarction within the last 6 months), congestive heart failure exceeding the New York heart association (NYHA) class III or IV, stroke, or transient ischemic attack.
9. Active clinical infection;
10. Symptomatic brain or meningeal metastasis (unless the patient is treated > At 6 months, imaging results were negative within 4 weeks prior to study entry and tumor-related clinical symptoms were stable at study entry);
11. Patients whose seizures require management (e.g. steroids or antiepileptic therapy);
12. Undergoing kidney dialysis;
13. Have a history of other malignant tumors within 3 years, except cured cervical carcinoma in situ or basal cell carcinoma of the skin;
14. Chronic intestinal diseases, infectious intestinal diseases, intestinal obstruction;
15. Drug abuse and medical, psychological or social conditions that may interfere with patient participation in the study or influence the evaluation of the study results;
16. Any unstable condition or condition that may compromise patient safety and poor compliance.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-08-31 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Sequential treatment of PFS with furoquitinib in second-line (F-C group) versus third-line (C-F group) | 10 months
  Sequential PFS is defined as:
  F-C group: time from randomization to disease progression or death after drug C, whichever occurred first.
  C-F group: time from randomization to disease progression or death after use of F drug, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Weijian Guo, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No